CLINICAL TRIAL: NCT07070440
Title: A Phase 1/2, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Efficacy of DZD6008 Combination Therapy in Patients With Locally Advanced or Metastatic NSCLC With EGFR Mutation (TIAN-SHAN7)
Brief Title: DZD6008 Combination Therapy in Patients With Locally Advanced or Metastatic NSCLC With EGFR Mutation (TIAN-SHAN7)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DZ2024C0001
Record Dates: First submitted 2025-06-16; First posted 2025-07-17 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DZD6008+pemetrexed/carboplatin (Experimental): DZD6008 was administered at 40/60/90 mg Once Daily (QD). Pemetrexed 500 mg/m2, once every 3 weeks, intravenous infusion. Carboplatin AUC 5 mg/mL/min, once every 3 weeks, intravenous infusion
  Interventions: Drug: DZD6008; Drug: Pemetrexed; Drug: Carboplatin
- DZD6008+docetaxel (Experimental): DZD6008 was administered at 40/60/90 mg QD. Docetaxel 75 mg/m2, once every 3 weeks, intravenous infusion
  Interventions: Drug: DZD6008; Drug: Docetaxel

INTERVENTIONS:
Drug: DZD6008 — DZD6008 was administered orally at 40/60/90 mg QD.
Drug: Pemetrexed — Pemetrexed 500 mg/m2, every 3 weeks, intravenous infusion.
  Arms: DZD6008+pemetrexed/carboplatin
Drug: Carboplatin — Carboplatin AUC 5 mg/mL/min, every 3 weeks, intravenous infusion.
  Arms: DZD6008+pemetrexed/carboplatin
Drug: Docetaxel — Docetaxel 75 mg/m2, every 3 weeks, intravenous infusion.
  Arms: DZD6008+docetaxel

SUMMARY:
This study is designed to evaluate safety and antitumor activity of DZD6008 combination therapy in patients with advanced Non-Small Cell Lung Cancer (NSCLC) with Epidermal Growth Factor Receptor (EGFR) mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age ≥18 years old.
3. Locally advanced or metastatic non-squamous non-small cell lung cancer by histopathology or cytology, not suitable for other radical treatment.
4. Documentation of EGFR sensitizing mutation confirmed by local laboratory.
5. Provide sufficient tumor tissue samples and plasma samples for retrospective analysis of EGFR mutations by central laboratory.
6. Failure of prior 3 generations EGFR TKI.
7. ECOG status score 0-1, life expectancy ≥12 weeks.
8. No central nervous system symptoms during screening, no need for corticosteroids or dehydration diuretic treatment for at least 4 weeks before the first dosing. If the patient with brain metastasis has received radiotherapy or surgery, there is a washout period of ≥2 weeks before the first use of DZD6008 and ensure that the AE related to radiotherapy or surgery has recovered to ≤ 1 grade.
9. Presence of measurable lesions defined by RECIST 1.1.
10. Sufficient bone marrow or other organ reserve before first dosing.

Exclusion criteria

1. Histology mixed with small cell lung cancer (SCLC) or with SCLC transformation.
2. Received the following treatments or had the following lifestyle habits, etc.:

   * Received immunotherapy or other antibody treatments (including EGFR-targeted antibodies, bispecific antibodies or antibody-drug conjugates, etc.) within 4 weeks before the first study drug administration.
   * Received any cytotoxic chemotherapy, study drugs or other anti-cancer drugs (excluding macromolecule drugs) within 14 days before the first study drug administration.
   * Received limited-range radiotherapy to relieve the disease within 7 days before the first study drug administration, or received more than 30% of the bone marrow radiotherapy or received wide-range radiotherapy within 28 days before the first medication.
   * 2 weeks (for CYP3A4 inhibitors) or 3 weeks (for CYP3A4 inducers) before the first study drug administration, are taking or cannot stop taking known cytochrome P450 (CYP) 3A4 strong inhibitors or inducers (including herbal supplements, such as St. John's wort).
   * 2 weeks before the first study drug administration, are taking or cannot stop taking known CYP3A4 sensitive substrate drugs (with a narrow therapeutic window).
   * Taking or being unable to stop taking drugs known to be proton pump inhibitors within 1 week before the first study drug administration.
   * Major invasive surgery has been performed within 4 weeks before the first study drug administration or is planned during treatment.
3. Presence of AEs of ≥1 grade (except any degree of alopecia) caused by previous treatment (such as adjuvant chemotherapy, radiotherapy).
4. Tumor-related spinal cord compression or meningeal metastasis.
5. History of malignant tumor within 2 years (except for basal cell carcinoma of the skin or cervical cancer in situ that has been adequately treated; other tumors that have been tumor-free for more than 2 years and are expected to survive for more than 2 years, which needs to be discussed with Dizal clinical research physicians).
6. Presence of severe or uncontrollable systemic diseases, including poorly controlled hypertension, bleeding diseases.
7. Presence of persistent or active infections, including but not limited to hepatitis B, hepatitis C and human immunodeficiency virus infection (HIV).
8. Any of the following heart-related diseases or abnormalities:

   * QT interval (QTc) >470 msec after calibration of 12-lead ECG at rest during the screening period.
   * Any serious abnormalities of heart rate, conduction or pattern shown on the ECG at rest, such as complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec.
   * Any disease or condition that can cause QTcF prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or family members with a history of sudden death under the age of 40.
   * Severe cardiovascular diseases such as myocardial infarction, unstable angina or congestive heart failure, cerebrovascular accident (such as history of stroke or intracranial hemorrhage) within 6 months before the first dose.
   * History of deep vein thrombosis or pulmonary embolism within 4 weeks before the first dose (excluding non-obstructive catheter-related thrombosis).
9. Patient history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid hormone treatment, or any clinically active ILD, immunotherapy-related pneumonitis.
10. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing medication, or previous intestinal resection that prevents adequate absorption of study medication.
11. Live vaccine within 4 weeks before the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose-limiting Toxicities (DLTs) | 21 days after the first dosing
  To assess safety and tolerability
Number of participants with Adverse events (AEs)/Serious adverse events (SAEs) | Through the study completion, an average of around 1 year.
  To assess safety and tolerability
Objective Response Rate (ORR) as assessed by investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Through the study completion, an average of around 1 year.
  To assess anti-tumor activity

SECONDARY OUTCOMES:
Duration of Response(DoR) | Through the study completion, an average of around 1 year.]
  DoR is defined as the time from the date of the first documented response (subsequently confirmed) according to RECIST 1.1 to the date of objective disease progression or death, whichever occurred first.
Disease Control Rate (DCR) | Through the study completion, an average of around 1 year.
  DCR is defined as the proportion of subjects with response defined as complete response, partial response, and stable disease according to RECIST 1.1 by the investigator.
Progression Free survival (PFS) | Through the study completion, an average of around 1 year.
  PFS is defined as the time from the first dose of the subject to objective disease progression based on RECIST 1.1 or death due to any cause (whichever occurs first).
Maximum Plasma/Serum Concentration (Cmax) of DZD6008 | Plasma samples were collected on day 1 of cycle 1, 2, 3, 5, 7, and 9, each cycle is 21 days
  Cmax = Maximum concentration
Time to Maximum Plasma/Serum Concentration (Tmax) of DZD6008 | Plasma samples were collected at cycle on day 1 of 1, 2, 3, 5, 7, and 9 , each cycle is 21 days
  Tmax = time to reach maximum concentration
Maximum Plasma/Serum Concentration (Cmax) of docetaxel | Plasma samples were collected on day 1 of cycle 1, 2, 3, 5, 7, and 9, each cycle is 21 days
  Cmax = Maximum concentration
Time to Maximum Plasma/Serum Concentration (Tmax) of docetaxel | Plasma samples were collected at cycles 1, 2, 3, 5, 7, and 9, each cycle is 21 days
  Tmax = time to reach maximum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Lu, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No